CLINICAL TRIAL: NCT04716725
Title: A Phase 2 Study of 68Ga-PSMA-11 PET in Patients With Metastatic Castration Resistant Prostate Cancer
Brief Title: 68Ga-PSMA-11 PET for the Diagnosis of Metastatic Castration Resistant Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Hope (Other)
Collaborators: Conquer Cancer Foundation (Other); Gateway for Cancer Research (Other); Prostate Cancer Foundation (Other)
Responsible Party: Sponsor-Investigator, Thomas Hope, Co-Principal Investigator (IND Holder), University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 209211; NCI-2020-13741 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-01-15; First posted 2021-01-20 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Castration-Resistant Prostate Carcinoma; Metastatic Prostate Carcinoma; Stage IV Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (68Ga-PSMA-11 PET) (Experimental): Patients receive gallium 68Ga-PSMA-11 IV and undergo PET at baseline, 16 weeks after initiating therapy, and at time of disease progression.
  Interventions: Drug: 68Ga-PSMA-11; Procedure: Positron Emission Tomography (PET)

INTERVENTIONS:
Drug: 68Ga-PSMA-11 — Given IV
  Other Names: 68Ga Prostate-specific Membrane Antigen (PSMA) 11; Gallium Ga-68 gozetotide; Gallium-68 PSMA; Gallium Ga 68 PSMA-11; Gallium Ga 68-labeled PSMA-11
Procedure: Positron Emission Tomography (PET) — Undergo PET
  Other Names: PET; PET Scan

SUMMARY:
This phase II trial studies the use of 68Ga-PSMA-11 positron emission tomography (PET) in diagnosing patients with prostate cancer that continues to grow despite the surgical removal of the testes or medical intervention to block androgen production (castration resistant), and has spread to other places in the body (metastatic). 68Ga- PSMA-11 is a new imaging agent that may help get more detailed pictures of the tumor. This trial aims to see whether using 68Ga-PSMA-11 PET scans may help doctors learn more about where disease is located in the body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether the percent change from baseline to 16 weeks (+/- 8 weeks) in maximum standard uptake value (SUVmax) averaged across up to 16 lesions per patient (SUVmax-ave) is associated with >= 50% decline from baseline in serum prostate specific antigen (PSA50) response.

SECONDARY OBJECTIVES:

I. To determine whether the percent change from baseline in SUVmax-ave on PSMA PET is associated with time-to-event endpoints including PSA progression-free survival and overall survival.

II. To determine whether the percent change from baseline in SUVmax on PSMA PET is associated with objective response by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 on a per-lesion basis among measurable soft tissue lesions present at baseline.

EXPLORATORY (CORRELATIVE) OBJECTIVES:

I. To descriptively characterize the histologic, transcriptional, and genomic features of PSMA low/negative lesions among patients who undergo paired optional metastatic tumor biopsy.

II. To descriptively characterize the relationship between SUVmax-ave on baseline Ga-PSMA PET with optional baseline fludeoxyglucose F-18 (FDG)-PET.

III. To determine whether heterogeneity of PSMA expression on baseline Ga-PSMA PET is associated with overall survival.

IV. To descriptively characterize the patterns of PSMA expression at the time of disease progression among patients who undergo optional PSMA PET.

V. To determine whether the percent change from baseline in PSMA PET is associated with PSA50 response among subgroups of patients defined by treatment modality received, including androgen receptor (AR) targeting treatment, PSMA-targeting radioligand therapy, cytotoxic chemotherapy, and immunotherapy.

OUTLINE:

Patients receive gallium Ga 68-PSMA-11 intravenously (IV) and undergo PET at baseline, 16 weeks after initiating therapy, and at time of disease progression.

After progression or study completion, patients are followed up every 3 months for up to 24 months

ELIGIBILITY:
Inclusion Criteria:

1. Sub-cohort A1: Patients must have baseline evaluations performed within 12 weeks prior to the start of systemic therapy.
2. Sub-cohort A2: Patients must meet all the following requirements:

   * Have had a baseline pre-treatment 68Ga-PSMA-11 PET scan and PSA measurement performed within 12 weeks prior to the start of current systemic therapy.
   * Able to have an on-treatment 68Ga-PSMA-11 PET and a PSA measurement within 16 weeks (+/- 8 weeks) after the start of current systemic therapy.

   Note: The screening period for sub-cohort A2 is within 24 weeks after the patient started their current systemic therapy.
3. Patients must have progressive castration resistant prostate cancer, according to PCWG3 criteria.
4. Patients must have planned initiation of systemic treatment (sub-cohort A1), or ongoing systemic treatment (sub-cohort A2) for castration resistant prostate cancer within 12 weeks of baseline Ga-PSMA PET.
5. Patients must have at least one metastatic lesion with PSMA uptake at or above the blood pool on their baseline PSMA PET scan.
6. The patient must be able and willing to comply with study procedures and provide signed and dated informed consent.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Patient must be Aged 18 years or older at the time of study entry.
9. Patients who undergo optional metastatic tumor biopsy following completion of baseline Ga-PSMA PET must additionally meet all of the following criteria:

   * Presence of one or more metastases by standard radiographic scans that is safely accessible to tumor biopsy in the judgment of treating clinician and/or Interventional Radiology.
   * No history of radiation therapy to the target metastatic lesion selected for tumor biopsy.
   * No contra-indication to biopsy including uncontrolled bleeding diathesis.
   * Platelets > 75,000/ul and prothrombin time (PT) or institution normalized ratio (INR) and a partial thromboplastin time (PTT) < 1.5 times the institutional upper limit of normal (ULN) within 14 days prior to biopsy.

Exclusion Criteria:

1. Patients who because of age, general medical or psychiatric condition, or physiologic status cannot give valid informed consent.
2. Patients with any condition that, in the opinion of the Principal Investigator, would impair the patient's ability to comply with study procedures.
3. Patients with any contra-indication to magnetic resonance imaging (MRI) (e.g. pacemaker placement, severe claustrophobia) Note: The exclusion criteria above (3) is only applicable for patients scheduled for a Positron Emission Tomography (PET) MRI (PET/MRI).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2025-04-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ivan A de Kouchovsky, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental (68Ga-PSMA-11 PET)
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental (68Ga-PSMA-11 PET)
Number analyzed (Participants) | 15
Age, Customized [Count of Participants; unit: Participants]
  40-49 years old | 1
  50-59 years old | 2
  60-69 years old | 2
  70-79 years old | 8
  80-89 years old | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Mean Maximum Standard Uptake Value (SUVmax)
Description: The mean SUVmax and standard deviation across the primary tumor and the 5 largest lesions in each of three metastatic sites (nodal, visceral and osseous; for a maximum of 16 lesions per patient) will be descriptively reported.
Time Frame: Baseline, and up to 16 weeks after initiation of therapy
Population: Data not collected
Arm/Group | Experimental (68Ga-PSMA-11 PET)
Number analyzed (Participants) | 0

2. Primary Outcome: Median SUVmax
Description: The median and range of SUVmax across the primary tumor and the 5 largest lesions in each of three metastatic sites (nodal, visceral and osseous; for a maximum of 16 lesions per patient) will be descriptively reported.
Time Frame: Baseline, and up to 16 weeks after initiation of therapy
Population: Data not collected
Groups:
- Experimental (68Ga-PSMA-11 PET): Participants receive gallium 68Ga-PSMA-11 IV and undergo PET at baseline, 16 weeks after initiating therapy, and at time of disease progression.
Arm/Group | Experimental (68Ga-PSMA-11 PET)
Number analyzed (Participants) | 0

3. Primary Outcome: Percentage of Participants Who Progressed by Prostate-specific Antigen (PSA) Response Group
Description: The percent of participants who fall into the PSA50 responders vs. non-responders based on PSMA treatment response criteria (PPP) for progression status will be reported. PPP uses 3 different criteria to determine response: 1) Appearance of 2 or more new PSMA positive distant lesions, 2) Appearance of 1 new PSMA positive lesion plus consistent clinical and/or laboratory data and recommended confirmation by biopsy or correlative imaging within 3 months of PSMA PET, and 3) Increase in size or PSMA uptake of 1 or more existing lesions by 30% plus consistent clinical and/or laboratory data and/or confirmation by biopsy or correlative imaging within 3 months of PSMA PET.
Time Frame: Baseline, and up to 16 weeks after initiation of therapy
Population: Participants were divided into subgroups based on whether or not the participant experienced a >= 50% decline from baseline in serum PSA
Measure: Number; unit: percentage of participants by group
Arm/Group | Experimental (68Ga-PSMA-11 PET)
Number analyzed (Participants) | 15
percentage of participants by group
  PSA Responders who progressed: number analyzed (Participants) | 9
  PSA Responders who progressed | 11.1
  PSA Non-Responders who progressed: number analyzed (Participants) | 6
  PSA Non-Responders who progressed | 83.3

4. Secondary Outcome: Comparison of Change in SUVmax-ave Group on Progression Free Survival (PFS)
Description: The study cohort will be dichotomized by the median with respect to percent change from baseline in SUVmax-ave on PSMA PET. The time-to-event variables including PSA progression-free will be defined by Prostate Cancer Clinical Trials Working Group 3 (PCWG3).
Time Frame: Up to 24 months
Reporting Status: Not Posted

5. Secondary Outcome: Comparison of Change in SUVmax-ave Group on Overall Survival (OS)
Description: The study cohort will be dichotomized by the median with respect to percent change from baseline in SUVmax-ave on PSMA PET on overall survival defined as time from imaging until death or censored at study completion. OS will be compared between dichotomized subgroups using the log-rank test. Kaplan-Meier product limit method will be used to estimate median survival in each subgroup.
Time Frame: Up to 24 months
Reporting Status: Not Posted

6. Secondary Outcome: Comparison Between Mean Percent Change in SUVmax With Objective Response Group
Description: Amongst the subset of measurable soft tissue lesions by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria, on a per-lesion basis, the mean percent change from baseline in SUVmax on PSMA PET will be compared between responding lesions defined as a complete response or partial response by RECIST 1.1 criteria vs. those without response, using Mann-Whitney test.
Time Frame: Baseline, and up to 16 weeks after initiation of therapy
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Experimental (68Ga-PSMA-11 PET)
All-Cause Mortality (participants affected / at risk) | 3/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

LIMITATIONS AND CAVEATS:
Participant enrollment closed earlier than anticipated due to slow accrual

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-08): https://cdn.clinicaltrials.gov/large-docs/25/NCT04716725/Prot_SAP_000.pdf